CLINICAL TRIAL: NCT01321281
Title: Randomised, Placebo Controlled Study to Determine if Aquamin (as AquaCal and AquaPT) Modulates Inflammatory Biomarkers in the Blood of Osteoarthritis and Healthy Subjects
Brief Title: A Study to Determine if Aquamin Modulates Inflammatory Biomarkers in the Blood of Osteoarthritis and Healthy Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Andrea Doolan (Other)
Responsible Party: Sponsor-Investigator, Andrea Doolan, Human Studies Manager, University College Cork
Organization: University College Cork (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: APC026-Marigot
Record Dates: First submitted 2011-03-22; First posted 2011-03-23 (Estimated); Last update posted 2012-05-15 (Estimated); Status verified 2012-05

CONDITIONS: Osteoarthritis
Keywords: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AquaCal (Experimental): Osteoarthritis and healthy volunteers
  Interventions: Dietary Supplement: AquaCal
- AquaPT (Active Comparator): Osteoarthritis
  Interventions: Dietary Supplement: AquaPT

INTERVENTIONS:
Dietary Supplement: AquaCal — AquaCal and AquaPT are produced by Marigot Ltd according to EU and FDA requirements.
  The daily dose of 4 capsules of AquaCal provide 800mg calcium, (the EU RDA for calcium) and 74 mgs Magnesium (EU RDA 375mg).
  Arms: AquaCal
Dietary Supplement: AquaPT — AquaCal and AquaPT are produced by Marigot Ltd according to EU and FDA requirements.
  The daily dose of 4 capsules of AquaPT provides 720mg calcium, 200mgs green tea (polyphenols) and 50 mgs pine bark extract.
  Arms: AquaPT

SUMMARY:
Osteoarthritis (OA) is the most common kind of arthritis and primarily affects the large, weight bearing joints (including the knees, lower back, hips, neck and the feet) and the joints in the hands. OA results from the breakdown of cartilage in joints, leading to joint pain and damage. It affects about 8 million people in the United Kingdom and nearly 27 million people in the United States, most of whom are over the age of 45.

This study aim to determine if Aquamin (as AquaCal and AquaPT) affects molecules of inflammation in the blood of osteoarthritis and healthy subjects.

DETAILED DESCRIPTION:
Aquamin is a seaweed-derived mineral source, which is rich in calcium, magnesium and 74 other trace minerals including zinc, iron and selenium. It is produced from the red algae, Lithothamnion Calcareum, which is found in just three locations in the world, including the south-west coast of Ireland and Iceland. During a five-year life span, these algae absorb essential minerals from the sea - this gives Aquamin its unique multimineral content. The algae then break down naturally and settle on the sea bed. These calcified skeletal remains are harvested, washed, dried and milled and provided in a capsule formulation. AquaCal is the capsule form of Aquamin. AquaPT contains green tea and pine bark extract.

Osteoarthritis (OA) is the most common kind of arthritis. OA is called degenerative arthritis, is a disease that results from the breakdown of cartilage in joints, leading to joint pain and damage. OA is very variable and there are lots of different types affecting different joints. This degenerative disease primarily affects the large, weight bearing joints (including the knees, lower back, hips, neck and the feet) and the joints in the hands. In OA, the disease begins with the degeneration of the cushion of cartilage between the joints. As it degrades, the synovium and the ends of the bones thicken, resulting in the pain and stiffness associated with arthritis. The progressive cartilage deterioration is followed by "hardening of the joints" due to calcification and bone spur formation. Treatment generally involves a combination of exercise, lifestyle modification and analgesics. If pain becomes debilitating joint replacement surgery may be used to improve the quality of life.

Symptoms of Osteoarthritis include early morning joint stiffness and pain, loss or restriction of joint mobility, pain that is worse after use, stiffness after periods of rest, creaking/cracking of joints after movement (also known as crepitus), tenderness and swelling in certain areas, restricted mobility, pain in the joint before or during changes in the weather and deformity of the joints.

Osteoarthritis is the leading cause of chronic disability in the United States.[1] It affects about 8 million people in the United Kingdom and nearly 27 million people in the United States, most of whom are over the age of 45. A number of studies have shown that there is a greater prevalence of the disease between siblings and especially identical twins, indicating a hereditary basis [2]. Up to 60% of OA cases are thought to result from genetic factors. Other factors causing OA are congenital disorders of joints, diabetes, inflammatory diseases and all chronic forms of arthritis. In addition, injury to joints as a result of an accident, septic arthritis, Marfan syndrome, obesity, ligamentous deterioration or instability may also be factors.

Current anti-inflammatory treatments for OA while providing some relief from symptoms are suboptimal and the side effects associated with these treatments; in particular the COX-2 specific NSAID's are becoming increasingly recognized [3,4]. As a result of this, use of alternative treatments and complementary medicines are gaining popularity among OA sufferers.

In a previous study, where osteoarthritis subjects were treated with Aquamin, there was a significant improvement in the WOMAC scores for pain, stiffness, activity and composite scores over the course of the 12-week treatment, in comparison to subjects in the Placebo group[5].

Aquamin is composed of multiple minerals and the 'active ingredient' for the complex is difficult to determine. A number of the minerals in Aquamin may have anti-inflammatory and anti-oxidant properties which might directly and/or indirectly influence the efficacy of this unique complex [7,8,9]. While the prominent mineral present in Aquamin is calcium (dosage = 80% Ca U.S RDA), its role in joint health is unclear. Magnesium however, was given at the daily dosage providing 14% (male) to 18% (female) U.S. RDA [6] and over the course of this study, this increased consumption of magnesium may have influenced OA symptoms by affecting the utilization of calcium or by potentially reducing inflammation around the affected joint. Both manganese and selenium were given at the daily dosage providing up to 16% and 4% of their RDA respectfully. Both of these trace minerals have been reported to reduce the appearance of osteoarthritic lesions and reduce the severity of symptoms in OA [8,9].

ELIGIBILITY:
Inclusion Criteria:

To be considered eligible for enrollment into the study, subjects must;

* Be able to give written informed consent.
* Be female and between 18 and 65 years of age.
* Be a non-pregnant female.
* Be in generally good health as determined by the investigator.
* Osteoarthritis patients must have a clinical diagnosis of moderate to severe osteoarthritis.

Exclusion Criteria:

Subjects will be excluded from the study if they meet any of the below criteria;

* Are less than 18 and greater than 65 years of age.
* Are pregnant females.
* Are currently taking probiotics or vitamin supplements, or have taken them in the past 14 days.
* Have a significant acute or chronic coexisting illness (cardiovascular, gastrointestinal, endocrinological, immunological, metabolic or any condition which contraindicates, in the investigators judgment, entry to the study).
* Having a condition or taking a medication that the investigator believes would interfere with the objectives of the study, pose a safety risk or confound the interpretation of the study results; to include non-steroidal anti-inflammatory drugs (NSAIDs), steroids and vitamin.
* Individuals who, in the opinion of the investigator, are considered to be poor attendees or unlikely for any reason to be able to comply with the trial.
* Subjects may not be receiving treatment involving experimental drugs.
* If the subject has been in a recent experimental trial, these must have been completed not less than 30 days prior to this study.
* Have a malignant disease or any concomitant end-stage organ disease.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2011-03; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Cytokines | Baseline (wk 0) & wk 6
  Plasma cytokine concentrations (including TNFα, IL-β, NFκB, COX2 & IL-6)

SECONDARY OUTCOMES:
WOMAC Questionnaire | Wk0 & Wk6
  Western Ontario and McMaster Universities Arthritis Index
Full Blood Count | Wk0 & Wk6
  Haemaglobin, white cell count, platelet count, haematocrit, differential white count
Chemistry Profile | Wk0 & Wk6
  Including Sodium, Potassium, Chloride, Urea, Creatinine, Protein, Albumin

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Dinan, Principal Investigator — University College Cork
Locations (1):
- Cork University Hospital, Cork, Ireland